CLINICAL TRIAL: NCT00884676
Title: A Phase I Trial of Weekly and Every Three Weeks Ixabepilone and Sunitinib in Solid Tumor Patients
Brief Title: Ixabepilone and Sunitinib Malate in Treating Patients With Progressive Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jaime Merchan (Other)
Collaborators: Bristol-Myers Squibb (Industry); Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Jaime Merchan, Associate Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20080376; GA6181ZB (Other Grant/Funding Number: Pfizer); CA163159 (Other Grant/Funding Number: Bristol Miers Squibb)
Record Dates: First submitted 2009-04-18; First posted 2009-04-21 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — ixabepilone; Sunitinib; Succinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Schedule A (Experimental): Schedule A: Ixabepilone - Weekly for 3 weeks each cycle (Days 1, 8 and 15) For both Schedules A and B, Sunitinib daily, orally, starting on Day 8 of Cycle 1
  Interventions: Drug: Ixabepilone; Drug: Sunitinib
- Schedule B (Experimental): Ixabepilone - Day 1 of each 3-week cycle For both Schedules A and B, Sunitinib daily, orally, starting on Day 8 of Cycle 1.
  Interventions: Drug: Ixabepilone; Drug: Sunitinib

INTERVENTIONS:
Drug: Ixabepilone — Administered intravenously. Dosage assigned by Phase I center as determined by dose-escalation schedule:
  * Schedule A: Weekly for 3 weeks each cycle (Days 1, 8 and 15)
  * Schedule B: Day 1 of each 3-week cycle.
  Other Names: BMS-247550; Ixempra; Azaepothilone B; epothilone B lactam; Epothilone-B BMS 247550
Drug: Sunitinib — For both Schedules A and B, daily, orally, starting on Day 8 of Cycle 1
  Other Names: Sunitinib Malate; Sutent; Butanedioic acid

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as ixabepilone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase I trial is studying the side effects and best dose of ixabepilone when given together with sunitinib malate in treating patients with progressive advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the safety and toxicity profile of ixabepilone in combination with sunitinib malate in patients with progressive, advanced non-hematologic malignancies.
* To determine the recommended phase II dose of ixabepilone given weekly versus once every three weeks in combination with a fixed dose of sunitinib malate in these patients.

Secondary

* To evaluate the pharmacokinetic profiles of the combination of ixabepilone and sunitinib malate and correlate them with activity and/or toxicity.
* To obtain preliminary efficacy data (complete response, partial response, or stable disease) of these treatment combinations.
* To correlate changes in angiogenesis biomarkers with clinical (safety and efficacy) and pharmacokinetic parameters in patients treated with these drug combinations.
* To estimate the optimal biological dose.

OUTLINE: This is a dose escalation study of ixabepilone. Patients are assigned to 1 of 2 treatment groups.

* Schedule A: Patients receive ixabepilone IV on days 1, 8, and 15. Beginning on day 8 of course 1, patients also receive oral sunitinib malate once daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
* Schedule B: Patients receive ixabepilone IV on day 1. Beginning on day 8 of course 1, patients also receive oral sunitinib malate once daily. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for biomarker and pharmacokinetic studies by flow cytometry.

After completion of study therapy, patients are followed at 30 days and every 3 months for 1 year.

ELIGIBILITY:
INCLUSION CRITERIA:

* Non-hematological malignancy that has progressed on standard therapy.
* Age > 18.
* ECOG Performance Status (PS) 0, 1, or 2.
* Life expectancy of > 3 months.
* More than three prior systemic therapy regimens (a period of 4 weeks from chemotherapy or immunotherapy ("washout period"), must have elapsed; and 2 weeks for prior tyrosine kinase inhibitors).
* Prior treatment with sunitinib in a 4 weeks on/2weeks off schedule is acceptable.
* Women of Child Bearing Potential (WOCBP) must use adequate method of contraception throughout and up to 4 weeks after the study.
* Patients must have either measurable disease (defined in Section 9.0) or evaluable disease (bony lesions, pleural effusion, ascites)
* Required laboratory values obtained <= 7 days prior to registration:

  * Granulocytes (ANC) >= 1500/mm3
  * PLT >= 100,000/mm3
  * Hgb >= 9.0 g/dL
  * Direct bilirubin <= 1.0 x ULN
  * Alkaline phosphatase <= 2.5 x ULN (<= 5 x if liver metastasis is present)
  * AST/ALT <= 2.5 x ULN (<= 5 x if liver metastasis is present)
  * Creatinine < 1.5 x ULN
  * Pregnancy Test Negative (For WOCBP*)
  * Urinalysis - Urine protein/creatinine ratio < 1, or < 1+ protein**
  * TSH = WNL
  * INR <= 1.5, unless the patient is on full dose warfarin or stable dose of LMW heparin with a therapeutic INR of > 1.5, <= 3.

    * Urine protein should be screened by random urine protein:creatinine ratio. For urine protein: creatinine ratio >1.0, 24-hour urine protein should be obtained and the level should be < 1000 mg for patient enrollment.
* Capable of understanding the investigational nature, potential risks and benefits of the study and able to provide valid informed consent.
* Willingness to donate blood for correlative marker studies.
* If a patient is on full-dose anticoagulants, the following criteria should be met for enrollment:
* The subject must have an in-range INR (usually between 2 and 3) on a stable dose of warfarin or on stable dose of LMW heparin.
* No active bleeding or pathological conditions that carry high risk of bleeding (e.g. tumor involving major vessels, known varices).

EXCLUSION CRITERIA:

* Patients with symptomatic/untreated CNS metastases. Patients with known CNS metastases can be enrolled if:
* CNS metastases have been appropriately treated. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, LINAC, or equivalent) or resection as deemed appropriate by the treating physician. Patients who had surgical resection of CNS metastases or brain biopsy within 3 months prior to Day 1 will be excluded.
* No ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period.
* No evidence of progression or hemorrhage after treatment (brain imaging study within 4 weeks of treatment start).
* CTC Grade 2 or greater neuropathy (motor or sensory) at study entry.
* Inability to swallow capsules.
* History of gastrointestinal disease, malabsorption, or requiring use of a feeding tube.
* Patients who have received any investigational compound within the past 28 days (within 2 weeks for prior RTKI treated patients).
* Patients who have received radiotherapy for any cause less than 4 weeks prior to study entry.
* Patients taking cytochrome P450 (CYP) 3A4 enzyme-inducing or enzyme-inhibitor medications like: antiepileptic drugs (phenytoin, carbamazepine or phenobarbital), St John's Wort, ketoconazole, dexamethasone, dysrhythmic drugs (terfenadine, quinidine, procainamide, sotalol, probucolol, bepridil, indapamide, or flecainide), haloperidol, risperidone, rifampin, grapefruit (or juice) within two weeks of registration and during the course of therapy. Topical and inhaled steroids are permitted. Please refer to Appendix VI for a complete list of CYP34A inducers and inhibitors.
* Patients with known HIV infection are excluded due to the possibility of unknown side effects on the immune system by these agents. The potential impact of pharmacokinetic interactions of anti-retroviral therapy with ixabepilone or sunitinib is unknown. Appropriate studies may be undertaken in patients with HIV and those receiving combination anti-retroviral therapy in the future.
* Invasive procedures defined as follows:

  * Major surgical procedure, open biopsy or significant traumatic injury <= 28 days prior to registration.
  * Anticipation of need for major surgical procedures during the course of the study.
  * Core biopsy <= 7 days prior to registration.
  * Port placement <= 7 days prior to registration.
  * Serious or non-healing wound, ulcer or bone fracture.
  * History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess <= 28 days.
* Evidence of bleeding diathesis or coagulopathy.
* Ongoing hemoptysis, or cerebrovascular accident <= previous 6 months, or peripheral vascular disease with claudication on < 1 block, or history of clinically significant bleeding.
* Significant cardiovascular disease defined as congestive heart failure (New York Heart Association Class II, III or IV), angina pectoris requiring nitrate therapy, or recent myocardial infarction (<= the last 6 months). Patients must have an absolute baseline left ventricular ejection fraction (LVEF) >= 50% by MUGA scan within 4 weeks prior to registration
* Uncontrolled hypertension (defined as a blood pressure of > 150 mmHg systolic and/or > 90 mmHg diastolic on medication).
* A currently active second malignancy other than non-melanoma skin cancer. Patients are not considered to have a currently active malignancy if they have completed anti-cancer therapy and are considered by their physician to be at less than 30% risk of relapse.
* Any of the following, as this regimen may be harmful to a developing fetus or nursing child:

  * Pregnant women
  * Breastfeeding women
  * Men or women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception (diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.) NOTE: The effects of the agent(s) on the developing human fetus at the recommended therapeutic dose are unknown.
* Other uncontrolled serious medical or psychiatric condition (e.g. cardiac arrhythmias, diabetes, etc.)
* Patients must not have ongoing ventricular cardiac dysrhythmias of NCI CTCAE Version 3.0 grade >= 2. Patients with a history of serious ventricular arrhythmia (VT or VF >= 3 beats in a row) are also excluded. Additionally, patients with ongoing atrial fibrillation are not eligible.
* Patients must have a QTc interval < 500 msec on baseline EKG.
* Prior treatment with ixabepilone.
* History of chronic or recurrent infection that requires continuous use of anti-viral, anti-fungal or anti-bacterial therapy; or foreseeable need to receive anti-infective therapy within 14 days of Cycle 1 Day 1 treatment.
* History of Grade 3/4 hypersensitivity reaction to Cremophor EL or its derivatives (polyoxyethylated castor oil).
* Non-small cell lung cancer (NSCLC) of squamous cell type, or NSCLC of any histology that involves a major blood vessel (e.g. aorta, pulmonary artery, etc)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-11; Primary Completion 2013-11 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Safety and toxicity profile as assessed by NCI CTCAE version 3.0 | Approximately 18-30 months
Recommended Phase II dose of Ixabepilone when administered with Sunitinib | Schedule A (12 - 18 months); Schedule B (6 -12 months after Schedule A)

SECONDARY OUTCOMES:
Pharmacokinetic profiles of Ixabepilone and Sunitinib malate and correlation with activity and/or toxicity | Approximately 18-30 months
Efficacy data (complete response, partial response, or stable disease) of these treatment combinations | Approximately 18-30 months
Correlation of changes in angiogenesis biomarkers with clinical (safety and efficacy) and pharmacokinetic parameters | Approximately 18-30 months
Estimation of optimal biological dose | Approximately 18-30 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaime R. Merchan, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida, United States